CLINICAL TRIAL: NCT07403318
Title: mHealth Supported Self-care Among Tertiary Education Students in Zimbabwe
Brief Title: Mobile Health Supported Self-care Among Tertiary Education Students in Zimbabwe
Acronym: MASCOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Centre for Sexual Health and HIV/AIDS Research Zimbabwe (CeSHHAR Zimbabwe) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MASCOT study; NIHR (Other Grant/Funding Number: NIHR303165)
Record Dates: First submitted 2026-01-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Unmet Need for Contraception; Uptake of HIV Prevention; Healthy Participants
Keywords: contraception; decision aid; young people; community-led; mHealth; adolescent girls and young women; adolescent boys and young men; HIV prevention; HIV post-exposure prophylaxis; HIV PEP; Emergency Contraception; peer-led interventions; student-led interventions

STUDY DESIGN:
Intervention Model Description: MASCOT is a suite of services that promote self-care among young people
  - using a peer-led model, supported by mobile health and decision aids to improve the uptake of HIV and contraception services. This multifaceted implementation strategy combines all three components of self-care in the following strategies: i) education - through peer distributors and through the mHealth tool. ii) decision support for a) HIV prevention, b) contraception - offered through decision aids, addressing self-awareness, potentially leading to self- management. iii) peer-led implementation - peers distributing self-care commodities (HIV self- test kits and condoms), and promoting self-care, addressing self-awareness, self-testing and self-management. Peer distributors will also promote and/ or refer students for additional HIV prevention services such as PEP, PrEP and voluntary medical male circumcision; and contraception services such as emergency contraceptive and other long acting contraceptive methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MASCOT intervention (Experimental): The MASCOT intervention is a suite of services that promotes self-care, using a peer-led model to distribute HIV and contraception services that is supported by a mobile health tool with decision aids. Students in the institutions where the MASCOT intervention is implemented will receive:
  1. education - through peer distributors and through the mHealth tool.
  2. decision support for a) HIV prevention, b) contraception - offered through decision aids, addressing self-awareness, potentially leading to self-management.
  3. peer-led implementation - peers distributing self-care commodities (HIV self-test kits and condoms), and promoting self-care, addressing self-awareness, self-testing and self-management. Peer distributors will also promote and/or referrals for additional HIV prevention services such as PEP, PrEP and voluntary medical male circumcision; and contraception services such as emergency contraceptive and other long acting contraceptive methods.
  Interventions: Other: MASCOT
- Standard of Care (No Intervention): Students in the standard of care arm will receive normal HIV prevention and contraception services.

INTERVENTIONS:
Other: MASCOT — A suite of services comprised of a peer-led model to deliver HIV prevention and contraception services using mobile health with decision aids to support self-care among students
  Arms: MASCOT intervention

SUMMARY:
Young people of ages 15-24 years, particularly those in Sub-Saharan Africa, do not optimally take up HIV services (HIV testing, HIV prevention and HIV treatment) and contraception. The number of new HIV infections in this group is disturbingly high and they suffer a lot of illness and death related to HIV. Research has found that four out of five sexually active adolescents in Africa are not using contraception. This means that millions of young people are exposed to unintended pregnancy and the associated negative effects such as unsafe abortions, school drop-out and reduced opportunities for both mother and baby. World Health Organisation have issued new guidelines for a new strategy, self-care, where an individual takes care of their own health and manages their illness with or without the support of a health worker. Self-care has potential to increase the number of young people who use HIV and contraception services. There is not enough information on how self-care can be done in a way that supports people to use services and maintain this use over time. Self-care can be made easier by mobile phone-based digital systems called mHealth, which may work by supporting access of services, for example where products are ordered online, or creating enabling conditions for self-care, for example through facilitating correct information-giving.

With various options for HIV prevention and contraception available, young people may need support/guidance choosing options that suit them. Health workers in overburdened health systems may be too overwhelmed to clearly present all options to guide informed decisions. Decision aids (tools that support patients/users to make informed choices that suit their values and preferences) can enhance self-care by enabling informed decisions. Decision aids for HIV prevention and contraception need to be developed for use in self-care settings. Combining decision aids with mHealth tools can enhance self-care.

This study will be co-developed with students enrolled in colleges/universities in Zimbabwe to develop a self-care strategy that includes mHealth together with decision aids and enables students to optimally use HIV and contraception services.

The study is divided into five stages, and builds on another study where a self-care strategy supported by an mHealth tool (without decision aids) was developed. In the first stage of the current study, preferences for decision aids and attributes to include in the mHealth tool will be obtained using qualitative research and a scoping literature review. In the second stage, findings from the first stage will be used to develop blueprints for two decision aids: one for contraception and the other for HIV prevention. In the third stage, the decision aids will be integrated with the existing mHealth tool through a crowdsourcing activity including students, and experts in health and mHealth. In the fourth stage the self-care strategy supported by mHealth and decision aids will be tested in a pilot at 2 colleges/universities. Finally, the fifth stage be a randomised control trial, across college/universities in Zimbabwe, to see whether the self-care strategy supported by mHealth and decision aids will be effective to promote self-care, and therefore, results in an increase in the uptake of HIV and contraception services. This study will also be applied to make recommendations on how the strategy can be provided outside of college/university contexts.

DETAILED DESCRIPTION:
Young people aged 15-24 years have the worst HIV and sexual and reproductive health outcomes of all ages globally. Across sub-Saharan Africa, only 65% of people living with HIV aged 15-24 years know their HIV status, compared with 84% of older adults. There is suboptimum uptake of condoms and other HIV prevention interventions, pre-exposure prophylaxis and voluntary medical male circumcision. Every week, 7,800 15-24 year olds are infected with HIV globally, of whom 25% are African women. More than 80% of sexually active adolescents in sub-Saharan Africa do not use contraception; millions of young people face unintended pregnancy, unsafe abortions and school drop-out.

Self-care, where an individual maintains their own health and copes with illness with or without health worker support, is a novel World Health Organisation (WHO)-recommended intervention that could increase uptake of services and achieve health targets. WHO recommends use of mHealth (using mobile devices such as mobile phones or other wireless technologies in medicine/ public health) to support self-care. Knowledge on how to most effectively implement and sustain self-care to optimise health outcomes is lacking. Rigorous evidence is needed to guide policy and practice.

This study will co-develop an empowering self-care intervention for young people, together with intended users. The self-care intervention aims to promote young people to take care of their own sexual and reproductive health through increasing uptake of HIV testing, prevention and care, and of contraception, with the ultimate goal of reducing HIV incidence and unintended pregnancies. The intervention will comprise self-care supported by innovative mHealth tools incorporating decision aids (tools that support patients/ users to make informed choices that suit their values and preferences) and digital support for continued engagement. The intervention builds on previous research on HIV self-testing, self-care, young people and mHealth.

Poor engagement in care and prevention is a huge public health challenge particularly among young people for whom the negative health and socio-economic consequences may persist for decades. Among young Africans living with HIV only 65% know their HIV status. In Zimbabwe, 50% and 34% of young men and women living with HIV have unsuppressed virus and young people with HIV have the highest mortality of any age group. Targets for voluntary medical male circumcision and pre-exposure prophylaxis have been missed and condom use has declined. HIV incidence is high; globally 28% of new HIV infections are among people aged 15-24 years. Demographic health surveys from 18 African countries found that 82.6% of sexually active 15-19-year- olds were not using contraception, with high rates of unintended pregnancies reported,5 exposing them to unsafe abortions, school drop-out and reduced opportunities for both mother and child.

Young people face many barriers to the uptake of HIV and sexual and reproductive health services. In addition, health services fail to support them to make informed decisions about the range of available options. Barriers to service uptake among young people include: fear of disclosure of HIV status/sexual activity, negative attitudes of health workers towards sexual activity in young people and lack of proximity to services. Poor knowledge and poor risk perception are also important: less than 50% of young Africans have comprehensive knowledge of HIV and 48% of those at high risk of infection perceive themselves to be at risk.

Self-care could empower individuals to engage in activities that promote health, prevent disease and manage illness by increasing patient choice, autonomy and access to services. Self-care was first recommended by WHO in 2019, with guidelines revised on a rolling basis according to emerging evidence.

Self-care includes three components:

i) self-awareness e.g. self-help, self-education, self-efficacy; ii) self-testing e.g. self-sampling, self-screening and self-diagnosis; iii) self-management e.g. self-treatment, self-examination.

A conceptual framework for self-care developed by Narasimhan and WHO has four domains. Central to self-care is upholding human rights, gender equality and other ethical values while taking a holistic patient-centred approach. Self-care can be accessed in various sites (home, community, pharmacies, health services, digital technologies). An enabling environment is critical (education/information, commodity security and supportive laws/policies) as is health system accountability: self-care should enhance health system reach rather than shift burden from health workers to patients.

Enhancing sexual and reproductive health among young people will influence their health and socio-economic outcomes for the rest of their life. This study has potential to curtail health and socio-economic challenges faced by young people now and in the future while reducing burdens on the over-stretched health systems in sub-Saharan Africa. Our research will provide evidence of potential public health impact versus costs and inform future scale-up of mHealth-supported self-care. mHealth solutions can effect positive behaviour change and improve quality and coverage of care. WHO recognises mHealth as important for achieving universal health coverage and recommends mHealth for self-care. mHealth technologies can support access e.g. ordering self-testing products or receiving results from self-collected samples. They can promote an enabling self-care environment where accurate information/education is disseminated. mHealth tools that link to health information systems enable documentation of use of services.

The topical study will incorporate decision aids for HIV prevention and contraception to support patient informed choices tailored to their values and preferences. For a health intervention with a choice of options, decision aids provide information on each option, including effectiveness, advantages, disadvantages and match with specified personal values/preferences. Few decision aids have been evaluated for HIV prevention, yet the growing number of prevention options (different formulations of pre-exposure prophylaxis - tablets, vaginal ring, injectable, formulations with/without contraception, in addition to other prevention options) mean that young people need decision support. Decision aids for contraception have been developed and are widely used; however, they will need adapting for African self-care contexts.

Importance of peer-led interventions The current study builds on a previous study that employed mHealth supported, peer-led delivery of HIV and sexual and reproductive health services among students enrolled in colleges/universities. Peer distribution of HIV commodities was found to be highly acceptable; and feasibility work found near universal uptake of HIV self-tests by peers. Preliminary work in the pilot shows high acceptability of peer-led self-care among students and supporting programs. Other studies have also reported on effectiveness of peer-led approaches among young people.

Research questions and aims The intervention to be co-developed and evaluated is called mHealth supported self-care among tertiary education students in Zimbabwe (MASCOT).

Research questions

1. How can the existing mHealth supported self-care package for HIV and sexual and reproductive be enhanced?
2. What is the impact of mHealth supported self-care on uptake of sexual and reproductive health services among college/university students in Zimbabwe?
3. What are the societal costs of mHealth supported self-care in Zimbabwe?
4. How can an mHealth supported self-care intervention co-developed with college/university students in Zimbabwe be adapted for youth in other settings? Aim: To determine how self-care can address the protracted challenge of poor service engagement among young people, with the ultimate goal of reducing HIV incidence and unintended pregnancies.

Specific objectives

1. Explore preferences for decision aids for HIV prevention and contraception and how decision aids can be incorporated into the existing self-care model among college/university students.
2. Adapt decision aids for HIV prevention and contraception for young people according to context-specific values and preferences
3. Adapt the existing mHealth tool to include support for decisions on uptake of HIV prevention and contraception.
4. Determine the feasibility and acceptability of MASCOT in two colleges/ universities
5. Determine effectiveness of MASCOT in improving uptake of HIV and contraception services and its societal costs in a cluster randomised trial in colleges/universities in Zimbabwe
6. Explore how MASCOT might be adapted for other settings through a detailed process evaluation Setting/context: The study will be conducted in Zimbabwean colleges/universities including technical colleges, teachers' training colleges, and so will capture a wide range of education abilities.

   Study overview

   Five work packages will drive this research:

   Work package 1 - Formative work to explore preferences for decision aids for HIV prevention and contraception and how to incorporate decision aids to the existing self-care intervention.

   Work package 2 - Development of decision aids for HIV prevention and contraception.

   Work package 3 - Using a hackathon to adapt the existing mHealth tool to include decision aids and a user interface Work package 4 - Pilot of mHealth supported self-care in two colleges/ universities.

   Work package 5 - Cluster randomised trial to determine the effect of mHealth supported self-care on uptake of HIV and contraception services.

   Description of the MASCOT intervention

   MASCOT uses a multifaceted implementation strategy combining all three components of self-care in the following strategies:

   i) Education or information-giving (addressing self-awareness) - through peer distributors and through the mHealth tool, overcoming poor knowledge.

   ii) Decision support for a) HIV prevention, b) contraception - offered through decision aids, addressing self-awareness, potentially leading to self-management. Overcomes challenges with informed decision-making.

   iii) Peer-led implementation - peers distributing self-care commodities and promoting self-care, addressing self-awareness, self-testing and self-management. Peers penetrate social circles, understand peer experiences and can package messages in understandable, acceptable ways.

   iv) Consumer and stakeholder involvement to ensure the intervention is acceptable and appropriate - students, Ministry of Health and other stakeholders involved in intervention design, implementation and evaluation, addressing self-awareness, self-testing and self- management.

   Conceptual Framework Intervention development is informed by the Narasimhan/WHO self- care framework and COM-B framework. COM-B specifies that three conditions are essential for behaviour change: capability, opportunity and motivation. MASCOT will enhance psychological capability by providing information through peer distributors and the mHealth tool including the decision aid. Physical capability will be enhanced by training/information giving on practical aspects of self-care (e.g. how to conduct HIV self-tests).

   MASCOT will address individual motivation to access contraception and/or HIV prevention/care by facilitating understanding of their risk through the decision aid. Self-care reduces the likelihood of deductive disclosure of sexual activity or HIV status by clinic staff or other clinic patrons - a major deterrent to service uptake. Widespread peer-driven implementation may also increase normalisation of self-care, potentially improving motivation.

   MASCOT will improve the opportunity to access contraception and HIV prevention/care through peer distribution of technologies and assisted access to clinical services for those who need them.

   Detailed study activities

   Work package 1 - Formative research

   Four to six focus group discussions with 8-12 participants each will be conducted among students aged 15-24 years to elicit values and preferences for HIV prevention and contraception decision aids and how they can be integrated to the existing self-care intervention. To help generate more informed views, students will interact with different examples of decision aids. Students will be purposively selected to include various disciplines, all gender and age groups, with representation across student years. Groups will be split by gender and age groups to encourage open/free participation. Key informant interviews will be held with 15-20 Ministry of Health officials and implementing partners to explore key attributes to be included in mHealth tools and decision aids. Qualitative studies will be conducted because they enable deep understanding of the explored phenomena. Interviews and focus group discussions will be analysed using a realist evaluation framework, targeting themes illustrating preferred attributes of mHealth tools and decision aids.

   Work package 2 - Developing decision aids

   Using findings from work package 1, a process to develop or adapt blueprints (detailed plans and content) of HIV prevention and contraception decision aids according to The International Patient Decision Aid Standards (IPDAS) will be conducted. The decision aids will be developed into electronic formats, following which, iterative testing will be done as part of work packages 3 and 4.

   Work package 3 - Adaptation of the parent mHealth tool

   Crowdsourcing, a process where a group of multi-disciplinary individuals solve a problem and solutions are shared with the public, will be applied to adapt the mHealth tool to include decision aids, user interface and additional preferences from Work package 1. One example of crowdsourcing is a hackathon where a group of people collectively solve a problem. In work package 3, a two- day hackathon will be held, bringing together different multi-disciplinary teams to compete against each other to adapt the parent mHealth tool to fit specifications defined in work packages 1 and 2. The hackathon will be organised according to WHO's practical guide for crowdsourcing. Finalists will be given prizes worth £2,000. The Implementation Advisory Committee will decide on the prize structure. Crowdsourcing was selected for tool development/adaptation because it allows systematic engagement of communities (potential users) with multi- disciplinary experts to formulate a product that is likely to have high user acceptance. It saves money compared to other digital tool development options, while generating an open-source product. There is evidence that crowdsourcing can result in high quality outcomes. The specifications of the required product will be provided, and judges (that include mHealth experts) will select the winning product. It is expected that the winning product will require considerable refinement to make it suitable for use; a technology development company will be engaged to complete development. The product will be tested iteratively among users and health workers before piloting in work package 4.

   Work Package 4 - Pilot of MASCOT intervention

   MASCOT will be implemented in two colleges/universities with a maximum enrolment of 3500 students each, to test the feasibility of MASCOT and data collection tools for measuring uptake, benefits and downsides (including burden on the health system). MASCOT will be implemented for six months followed by a survey conducted among 15% of enrolled students to measure uptake of HIV and sexual and reproductive health services.

   A detailed process evaluation, using mixed methods will be done according to the realist evaluation framework. The process evaluation will explore how context shapes implementation, fidelity to implementation, and perceptions of what works well and less well. It will involve i) analysis of program data on uptake of various self-care components, linkage and/or retention, ii) qualitative in-depth interviews with students who interacted with MASCOT and those who have not. Detailed costing of MASCOT will also be done. Pilot findings will be used to refine the MASCOT intervention, data collection tools, randomisation and primary outcomes (detailed below in work package 5).

   Work Package 5 - Cluster randomised trial

   A cluster randomised trial will be conducted in 24 colleges randomised 1:1 to MASCOT or standard of care. Randomisation will be restricted by college/university size, female/male ratio, and college type. Colleges will be selected across ten provinces in Zimbabwe, and will be geographically separated by at least 20km to prevent contamination. In intervention colleges the MASCOT intervention will be implemented for six months. Baseline and endline representative in-person surveys will be conducted among 15% of students that are randomly selected. The students will self-complete the survey questionnaire on tablets. Additionally, dried blood spot samples will be collected for HIV testing, and for those testing HIV-positive, viral load tests will also be performed. All students enrolled at the colleges/universities for at least 6 months and willing to provide informed consent for the survey will be eligible to participate, regardless of whether they participated in MASCOT. Detailed process evaluation will be conducted as in work package 4.

   Detailed costing of MASCOT will be done from the societal perspective, using standard methods for cost analysis to capture both provider and user costs. Program costs will be collected using a costing tool. Information on program start up and implementation will be collected for costing analyses. Care will be taken to include the costs incurred by peer distributors in intervention implementation, including in-kind costs. Costs of accessing services will be estimated using costing surveys among students. Peer distributors will be trained to collect cost data, thus building their capacity for costing community-led interventions.

   Impact of study

   This study will produce evidence on how self-care can be implemented among college students in Southern Africa, with recommendations for adaption for other contexts. Outputs will include an open access, context-relevant mHealth tool with decision aids for HIV prevention and contraception.

ELIGIBILITY:
Work package 1: Formative research

1. Focus Group Discussions

   * Aged 16 years old or over;
   * Currently enrolled at a college/university where the research is being done;
   * Willing and able to provide written informed consent.

   Exclusion Criteria:

   - None stated
2. Key informant interviews

   * Staff from MoHCC responsible for implementing or supervising implementation of HIV or sexual and reproductive health services, or for policy planning on the same topics,
   * Staff from Ministry of Higher and Tertiary Education responsible for student health, staff from Ministry of Health implementing partners working on HIV and sexual and reproductive health services in Zimbabwe,
   * Willing and able to provide written informed consent.

Exclusion Criteria:

- None stated

Work package 3: Adaptation of the parent mHealth tool

1. Hackathon

1a. Students

Inclusion criteria:

* Enrolled in the specific institutions; in these disciplines: public health, information technology and computer science; and
* Willing to take part in the hackathon

Exclusion criteria:

None stated

1b. Multi-disciplinary experts

Inclusion criteria:

* Representatives in any of the following disciplines, Digital health experts, MoHCC, HIV and SRH services, other key stakeholders; and
* Willing to take part in the hackathon.

Exclusion criteria:

None stated

2. Alpha testing

2a. Students

Inclusion criteria:

• Recruited from the same colleges/universities that participated in formative research

• Willing and able to provide written informed consent.

Exclusion criteria:

None stated

2b. Health workers

Inclusion criteria:

* Staff from MoHCC responsible for implementing or supervising the implementation of HIV and sexual and reproductive health services,
* Willing and able to provide written informed consent.

Exclusion criteria:

None stated

3. Beta testing

3a. Students

Inclusion criteria:

* Students who have used the mHealth tool and decision aids
* Willing and able to provide written informed consent.

Exclusion Criteria:

- None stated

4. Pilot of mHealth supported self-care in two colleges/universities

4a. Institutions

Inclusion criteria:

* Less than 3500 students
* Comparable male and female ratio
* Participated in formative research

Exclusion criteria:

Institutions that participated in the formative research

4b. Peer distributors

Inclusion criteria:

* Aged >18 years;
* Currently enrolled at the participating colleges/universities
* Willing to be a peer distributor,
* Willing to conduct study activities according to the protocol.

Exclusion criteria:

- Students who were away from college for industrial attachment during intervention implementation

4c. Pilot survey

Inclusion criteria:

* Students enrolled at the colleges/universities for at least 6 months.
* Willing to provide written informed consent for the survey.

Exclusion criteria:

- Students who were away from college for industrial attachment during intervention implementation

4d. In-depth interviews with students

Inclusion criteria:

* Students enrolled at the colleges/universities for at least 6 months.
* Willing to provide written informed consent for the in-depth interviews

Exclusion criteria:

None defined

4e. In depth interviews with Peer Distributors

Inclusion Criteria:

* Student peer distributor at a tertiary education institution where the research is being done; and
* Willing and able to provide written consent for the interview.

Exclusion criteria:

None defined

4f. FGDs with students

Inclusion criteria:

* Enrolled at the colleges/universities for at least 6 months.
* Willing to provide informed consent for the FGD.

Exclusion criteria:

None defined

4g. In depth interviews with health workers

* Health worker at participating college/university supporting the MASCOT intervention.
* Willing and able to provide written informed consent.

Exclusion criteria:

None defined

5. Cluster Randomised trial

5a. Institutions

Inclusion criteria:

* Located in 10 provinces: Harare, Mashonaland Central, West and East, Masvingo, Manicaland, Midlands Bulawayo and Matabeleland North and South
* Maximum enrolment of 3500 students

Exclusion criteria:

None defined

5b. Surveys, in-depth interviews with students, peer distributors and health workers and FDGs with students will be the same as for work package 4 above.

5c. Costing interviews with distributors

Inclusion criteria:

* Student peer distributor at a tertiary education institution where the research is being done; and
* Willing and able to provide written consent for the costing interview.

Exclusion criteria:

None defined

5d. Costing - Valuing distributor time

Inclusion criteria:

* Student peer distributor at a tertiary institution where the research is being done.
* Willing and able to provide written consent

Exclusion criteria:

None defined

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16000 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of students at risk of HIV acquisition | At the end of implementation of MASCOT, at 6 months
  In work package 5, a cluster randomised control trial will be conducted at colleges/universities to compare the effectiveness of MASCOT in promoting uptake of HIV and sexual and reproductive health services among young people in colleges/universities. After six months of implementing MASCOT, a population representative survey will be conducted among 15% of randomly selected students attending participating colleges/universities, regardless of interacting with MASCOT. This survey will include collection of dried blood spots from participants, for HIV testing and in HIV-positive samples, viral load testing.
  The numerator for this outcome is: total number of students at risk of acquiring HIV, defined as: HIV negative students (obtained from HIV negative result from blood spot testing) that are engaging in risky sex and not using HIV prevention methods (self-reported based on survey response).
  The denominator for this outcome is: the total number of surveyed students.
Proportion of students using effective contraception | At the end of implementation of MASCOT, at 6 months
  In work package 5, a cluster randomised control trial will be conducted at colleges/universities to compare the effectiveness of MASCOT in promoting uptake of HIV and sexual and reproductive health services among young people in colleges/universities. After six months of implementing MASCOT, a population representative survey will be conducted among 15% of randomly selected students attending participating colleges/universities, regardless of interacting with MASCOT. This survey will include questions on contraception use.
  The numerator for this outcome is: total number of students using effective contraception when having sex with a partner measured (self-reported based on survey responses).
  The denominator for this outcome is: total number of surveyed students.

SECONDARY OUTCOMES:
Provider and societal cost per contraceptive/HIV service taken up | From study inception to the end of implementation of intervention at 6 months
  Trained economics data collectors including peer distributors will use a specially designed costing tool to collect information on activities contributing to program roll-out. The tool will record data on preparatory activities such as community entry and engagement workshops with key relevant stakeholders, value program and distributor (personnel) time, MASCOT commodities, vehicle and travel and other recurrent costs.
  For students, accessing HIV prevention and contraception services may involve travel (e.g., to collect EC or get confirmatory testing) and other costs in addition to productivity losses, which may potentially deter uptake. We will therefore aim to characterize these costs of accessing services in work package 5 post-intervention representative in-person surveys which will be conducted among 15% randomly selected students in each trial college. Only selected students who answer yes to accessing all or any MASCOT commodities will be included.
Proportion of students at risk of HIV transmission | At the end of study implementation, at 6 months
  In work package 5, a cluster randomised control trial will be conducted at colleges/universities to compare the effectiveness of MASCOT in promoting uptake of HIV and sexual and reproductive health services among young people in colleges/universities. After six months of implementing MASCOT, a population representative survey will be conducted among 15% of randomly selected students attending participating colleges/universities, regardless of interacting with MASCOT. This survey will include collection of dried blood spots from participants, for HIV testing and viral loading. The numerator for this outcome is: total number of students at risk of transmitting HIV, defined as: HIV positive students who are not virally suppressed (obtained from blood testing).
  The denominator for this outcome is: total number of surveyed students.
Quantitative implementation outcomes | From enrollment to the end of implementation at 6 months
  Based on program data: 1) numbers taking up each of the self-care services 2) numbers interacting with the decision aids. These data will be collected through the mHealth tool.
Qualitative implementation outcomes - Feasibility, acceptability, fidelity and impact of the study. | From enrollment to the end of implementation at 6 months
  Feasibility- Qualitative studies will be used to assess whether MASCOT can be effectively implemented in practice. Feasibility will also be measured by analysing program data on: uptake of commodities (through mHealth tool), and use of decision aids (through mHealth tool).
  Acceptability- Qualitative interviews will be used to assess how well MASCOT was received by the target population and stakeholders. Program data (from mHealth tool) will be collected to determine acceptability of MASCOT.
  Fidelity- Qualitative interviews will be used to assess the degree to which the MASCOT intervention was implemented as intended or designed. Fidelity will be assessed on adherence to the peer-led model and mHealth use to promote uptake of HIV/SRH services.
  Impact- We will also use qualitative interviews to assess broader changes that may occur because of MASCOT over time. Data will be collected on potential contribution of MASCOT to improve uptake of HIV and contraception services.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Sexual Health and HIV/AIDS Research Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code